CLINICAL TRIAL: NCT01144273
Title: Transversus Abdominis Plane Block From Intraabdominal Approach in Patients Undergoing Total Abdominal Hysterectomy: a Randomized Controlled Trial
Brief Title: Transversus Abdominis Plane Block From Abdominal Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United Christian Hospital (Other)
Responsible Party: Dr Choy Wing Yee Lillian, United Christian Hospital, Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Protocol ver 1.1; KC/KE-10-0021/FR-3 (Other: Research Ethics committee (Kowloon Central/Kowloon East))
Record Dates: First submitted 2010-06-14; First posted 2010-06-15 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Transversus Abdominis Plane Block From Abdominal Approach

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5% Ropivacaine (Active Comparator): group receiving TAP block (0.5% ropivacaine at TAP plane)
  Interventions: Procedure: Transversus abdominis plane block
- normal saline (Placebo Comparator): group receiving placebo (saline) at TAP plane
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — This intraabdominal approach to TAP block is being used regularly by gynaecological surgeons in this hospital now.
  To be performed bilaterally before surgical wound closure by an experienced surgeon who initially undergo initial observation by investigator to ensure uniformity in technique.
  Local anaesthetic or placebo solution will be injected to TAP with blunt needle from within abdominal cavity under visual and tactile guidance at the triangle of Petit, after feeling one 'pop' through the transversus abdominis muscle to the TAP layer.
  After careful aspiration to exclude vascular puncture, 1.5mg/kg of 0.5% ropivacaine or 0.3ml/kg of 0.9% saline placebo will be injected to each side slowly while observing for signs of toxicity.
  Other Names: TAP block

SUMMARY:
Randomized double blind placebo controlled trial on transversus abdominus plane block approached from abdominal cavity, in patients undergoing total abdominal hysterectomy.

DETAILED DESCRIPTION:
Potential advantages compared to percutaneous approach are decrease in risk of visceral injury as it is under direct visual and tactile guidance, ease of approach in obese patients, short theatre time for administration, easy to administer.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-III
* Age 18 or above
* Scheduled to undergo TAH+/- salpingoophorectomy.
* Scheduled to receive general anaesthesia under standardized anaesthetic regime.
* Comprehends how to use intravenous patient controlled analgesia (IV PCA).
* Is willing to complete the postoperative assessment.
* Understands the nature and purpose of this study and the study procedures and has signed the informed consent form for this study to indicate this understanding.

Exclusion Criteria:

* Known allergy to drugs involved in this study
* Previously taking medications thought to result in opioid tolerance, or analgesics thought to interfere with subsequent opioid requirement.
* Undergoing any procedures in addition to TAH+/- salpingoophorectomy.
* With co-existing pathology resulting in persistent pain requiring analgesics.
* Wound incision extending to supra-umbilical level.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
postoperative 24hr morphine consumption | 24 hours
  The primary objective of this study is to demonstrate the effectiveness of tranversus abdominis plane block using the intraabdominal approach in reducing postoperative 24 hours morphine consumption after total abdominal hysterectomy (TAH) where time 0 is taken as time of arrival at PACU.

SECONDARY OUTCOMES:
morphine consumption on arrival to post-anaesthetic care unit(PACU) and 4, 12 and 24 hours after. | 24hrs
  • Assess and compare the morphine consumption on arrival to post-anaesthetic care unit(PACU) and 4, 12 and 24 hours after.
Degree on pain according to numerical pain score on arrival to post-anaesthetic care unit(PACU) and 4, 12 and 24 hours after during rest and movement (cough | 24hrs
incidence of nausea and vomiting | 24hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Wing Yee Lillian Choy, MBBS (HK), Principal Investigator — United Christian Hospital, Hospital Authority
Locations (1):
- Department Of Anaesthesiology, Pain medicine and Operating Services. United Christian Hospital, Kwun Tong, Kowloon, Hong Kong

REFERENCES:
- [Background] McDonnell JG, O'Donnell B, Curley G, Heffernan A, Power C, Laffey JG. The analgesic efficacy of transversus abdominis plane block after abdominal surgery: a prospective randomized controlled trial. Anesth Analg. 2007 Jan;104(1):193-7. doi: 10.1213/01.ane.0000250223.49963.0f. PMID 17179269
- [Background] Carney J, McDonnell JG, Ochana A, Bhinder R, Laffey JG. The transversus abdominis plane block provides effective postoperative analgesia in patients undergoing total abdominal hysterectomy. Anesth Analg. 2008 Dec;107(6):2056-60. doi: 10.1213/ane.0b013e3181871313. PMID 19020158
- [Background] Bonnet F, Berger J, Aveline C. Transversus abdominis plane block: what is its role in postoperative analgesia? Br J Anaesth. 2009 Oct;103(4):468-70. doi: 10.1093/bja/aep243. No abstract available. PMID 19749115